CLINICAL TRIAL: NCT00609921
Title: A Phase 1 Dose Escalation Study of ARQ 197 in Adult Patients With Advanced/Recurrent Solid Tumors
Brief Title: A Phase 1 Study of ARQ 197 in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARQ 197-0701
Record Dates: First submitted 2008-01-25; First posted 2008-02-07 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-09

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — ARQ 197

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Active Comparator): ARQ197
  Interventions: Drug: ARQ197

INTERVENTIONS:
Drug: ARQ197 — treatment

SUMMARY:
This is a Phase 1, open label, dose escalation study of ARQ 197 in patients with advanced/recurrent solid tumors. The purpose of this study is to determine the safety, tolerability and recommended Phase 2 dose (RP2D) of ARQ 197.

ELIGIBILITY:
Inclusion Criteria:

* Patients who did not respond or are refractory to available therapy or for whom no standard effective systemic therapy exists.
* Karnofsky performance status (KPS) ≥ 70%, or Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1
* Patients with adequate organ function

Exclusion Criteria:

* Anti-cancer chemotherapy, hormonal therapy, radiotherapy, immunotherapy, or investigational agents within 4 weeks prior to the first dose of ARQ 197
* Known symptomatic brain metastases
* Pregnant or breastfeeding
* Uncontrolled intercurrent illness

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2008-01; Primary Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Determine the safety, tolerability and recommended Phase 2 dose (RP2D) of ARQ 197

SECONDARY OUTCOMES:
Assess the preliminary anti-tumor activity and determine the pharmacokinetic profile

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Kyowa Kirin Co., Ltd.